CLINICAL TRIAL: NCT03734510
Title: Evaluation of the Effects of Supplementation of Flaxseed, Hesperidin, Flaxseed and Hesperidin Together on Hepatic Enzymes, Inflammatory Factors, Lipid Profile, Blood Glucose, Insulin Sensitivity, and Hepatic Steatosis Grade in Patients With Non-alcoholic Fatty Liver Disease
Brief Title: The Effect of Supplementation of Flaxseed, Hesperidin, Flaxseed and Hesperidin Together in Non-alcoholic Fatty Liver Disease: A Randomized, Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, MD, PhD, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13679
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Linseed Oil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- hesperidin and flaxseed (Active Comparator)
  Interventions: Dietary Supplement: Dietary Supplement: hesperidin and flaxseed
- control (Placebo Comparator)
  Interventions: Other: control
- flaxseed (Active Comparator)
  Interventions: Dietary Supplement: Dietary Supplement: flaxseed
- hesperidin (Active Comparator)
  Interventions: Dietary Supplement: Dietary Supplement: hesperidin

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: hesperidin and flaxseed — 2 capsules hesperidin and 30 g flaxseed
  Arms: hesperidin and flaxseed
Dietary Supplement: Dietary Supplement: hesperidin — 2 capsules hesperidin
  Arms: hesperidin
Dietary Supplement: Dietary Supplement: flaxseed — 30 g flaxseed
  Arms: flaxseed
Other: control — no supplementation
  Arms: control

SUMMARY:
To study the effects of Hesperidin, flaxseed and both together on lipid profile, liver enzymes, inflammatory factors and hepatic fibrosis in patients with Nonalcoholic Steatohepatitis (NASH), 100 patients who referred to Gastrointestinal (GI) clinic with steatosis grade 2 and 3 will be randomly allocated to one of following four groups: control group, hesperidin group (2 capsules Hesperidin), flaxseed group (30 gram flaxseed) or flaxseed-hesperidin group (2 capsules Hesperidin and 30 gram flaxseed) for 12 weeks; both groups will be advised to adherence the investigators' diet and exercise program too. At the first and the end of the intervention, lipid profiles, liver enzymes, some inflammatory markers, and liver fibrosis will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 70 years
* Body Mass Index (BMI) between 25-40
* Sonographic findings compatible with hepatic steatosis (degree 2 or more)

Exclusion Criteria:

Diabetes Taking any kind of antibiotics two weeks before recruitment History of alcohol consumption pregnancy or lactation Professional athletes Other liver disease (viral/etc) Use of drugs such as calcium channel blockers, high dose synthetic estrogens, methotrexate , amiodarone, steroids, chloroquine, immunosuppressive drugs, lipid-lowering agents, metformin and vitamin E A history of Hypertension, Cardiovascular disease, Pulmonary disease, Renal disease & Celiac disease; Cirrhosis History of Upper GI surgery / Prior surgical procedures such as jejunoileal or jejunocolic bypass, gastroplasty Following program to lose weight in recent 3 mo A history of hypothyroidism or Cushing's syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
liver fibrosis | 12 weeks
  assess by fibroscan

CONTACTS AND LOCATIONS:
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran (the Islamic Republic Of), Iran